CLINICAL TRIAL: NCT06700642
Title: The Impact of Individual Education on Rational Drug Use in Primary Care for Patients on Long-Term Medication: an Intervention Study
Brief Title: Individual Education on Rational Drug Use in Primary Healthcare for Patients on Long-Term Medication
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gülşah Onur (Other)
Responsible Party: Sponsor-Investigator, Gülşah Onur, Research Assistant Dr., Hacettepe University
Organization: Hacettepe University (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: HUTF-FM-GODAB-01
Record Dates: First submitted 2024-11-20; First posted 2024-11-22 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-11

CONDITIONS: Medication Adherence; Patient Compliance; Drug Utilization Review
Keywords: family practice; rational drug use; medication adherence; controlled clinical trials; aging; noncommunicable diseases
MeSH Terms: conditions — Medication Adherence; Patient Compliance; Noncommunicable Diseases | interventions — Early Intervention, Educational

STUDY DESIGN:
Intervention Model Description: In the design of the study, in order to fix the effect of possible confounding variables for the research and control arms, 36 groups formed according to the distribution of gender, age groups and education levels of the research arm were matched to the control arm in terms of these characteristics.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Research Arm (Active Comparator): Individuals in this arm were given individual education on rational drug use by the researcher at the first visit. 'Individual Training Presentation on Rational Drug Use' consisting of visual and written content was used for patient education intervention. After the education, 'Rational Drug Use Patient Brochure' was given to all participants in this arm.
  Interventions: Other: Educational intervention
- Control Arm (No Intervention): No educational intervention was made in the control arm and no brochure was given at the first visit. In line with the principle of equality, participants in this arm were given a patient brochure at the end of the study.

INTERVENTIONS:
Other: Educational intervention — In this study, 3 intervention tools were developed by the researchers. The first of these, 'Rational Drug Use Trainer Guide', was used for trainer training and standardisation of the education given to patients. The sample rational drug use presentations prepared by the Ministry of Health, Turkiye Medicines and Medical Devices Agency, Department of Rational Drug Use were combined in terms of content, enriched with information obtained from the literature and developed for the use of family physicians working in primary health care institutions in their clinical practices.
  'Rational Drug Use Individual Education Presentation' was prepared by the researchers in line with the 'Rational Drug Use Trainer Guide'. It has been prepared in a format suitable for individual education presentation with the most concise and understandable content suitable for use during primary healthcare service delivery.
  'Rational Drug Use Patient Brochure' was prepared by the researchers in a similar content.
  Arms: Research Arm

SUMMARY:
Irrational medication use is a common problem in Turkiye and worldwide. Educational interventions are essential to promote rational drug use. This study was conducted to evaluate the effect of individual education on rational drug use given to individuals aged 45-74 years with at least one continuously used medication who applied to a primary health care institution on their rational drug use level. The hypothesis of the study was that individual training on rational drug use given to individuals using medication continuously is effective in increasing rational drug use.

DETAILED DESCRIPTION:
Incorrect, unnecessary, ineffective and high-cost drug use is a significant problem all over the world. The adherence of patients to the treatment recommended by the healthcare professional depends on the improvement of their knowledge, attitudes and behaviours about rational drug use (RDU) in the correct direction. There is a need for educational interventions that will increase the knowledge and awareness of the society on this matter and encourage RDU. This study was conducted in Hacettepe University Faculty of Medicine, Family Medicine Training Unit to evaluate the effect of RDU education in individuals aged 45-74 years who were continuously taking medication. In this non-randomised matched controlled intervention study, participants who met the criteria were non-randomly divided into two groups (research and control arm). Firstly, volunteers for the research arm started to be included in the study. According to the distribution of gender, age groups and education levels of the research arm, a one-to-one matching was made to the control arm in terms of these qualifications. In this way, the effects of three possible confounding variables for the two arms were controlled through group matching. In the first visit, data were collected from the research and control arms with questionnaire forms including sociodemographic information and the Rational Drug Use Scale (RDUS). In the first visit after the completion of the questionnaire form, each individual in the research arm was given individual-patient education on rational drug use and patient brochure by the researcher. The control arm received no educational intervention and was not given a brochure at the first visit. The final visit was conducted with both the research and control arms 3 months after the first visit of each individual. The effect of the educational intervention on RDU was evaluated with the RDUS. In this visit, the individuals in the control arm were also given a patient brochure in line with the 'principle of equality'.

ELIGIBILITY:
Inclusion Criteria:

* Taking at least one medication continuously (Individuals with taking at least one medication that 'has been used every day for a minimum of 3 months and should be used for at least 1 year' were defined as 'continuous medication users'. Patients' declarations of continuous medication use were verified through the Family Medicine Information System).
* To be between 45-74 years old
* Not being dependent on another individual in terms of medication use
* Being co-operative and orientated (The Mini Mental Test is routinely administered to individuals over the age of 65 who are registered in the Family Medicine Training Unit and the results of this test can be seen in the Family Medicine Information System. In our study, those with normal scores (between 24-30 points) were considered to be co-operative and orientated).
* To be at least primary school graduate
* To agree to participate in the study

Exclusion Criteria:

* Not to have a medication that is used continuously
* Under 45 years of age or 75 years of age or older
* Being a cancer patient in active treatment
* Being pregnant or breastfeeding
* Having a severe psychiatric disorder
* Uncooperative or disorientated
* Not having completed primary school education
* Getting help from another person for the use of medicines
* In the recruitment of volunteers for the control arm to the 36 groups formed according to the distribution of gender, age groups and education levels of the research arm, the absence of a participant suitable for the characteristics of the group (In order to stabilise the effect of possible confounding variables between the two arms, each participant in the research arm was matched one-to-one with the participants in the control arm in terms of three sociodemographic variables. In the recruitment of volunteers to the control arm, if there was no participant matched to the age group, gender and education level of the participant in the research arm, the participants who were last included in the study in the research arm and could not be matched were excluded from the study).
* Development of a medical condition that prevented participation in the final visit within the three-month follow-up period

Ages: 45 Years to 74 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 365 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2024-01-12 (Actual); Study Completion 2024-04-16 (Actual)

PRIMARY OUTCOMES:
The effect of individual education on rational drug use status | 3 months after the first visit of each individual with both the research and control arm
  Rational drug use status of the participants was measured with the Rational Drug Use Scale (RDUS). The RDUS consists of 21 questions and a single dimension. In this 5-point Likert-type scale, the answers for each item are never (1 point), rarely (2 points), sometimes (3 points), often (4 points) and always (5 points). Only the 17th item in the scale is reverse scored. After the reverse scoring process, the 'total scale score' is calculated by summing the scores of all items of the scale. As the total score obtained from RDUS increases, rational drug use also increases.
  This scale was applied to both arms in both first visit and final visit, and the effect of the educational intervention was evaluated through this scale.

CONTACTS AND LOCATIONS:
Overall Officials: Gülşah Onur, Research Assistant Dr., Principal Investigator — Hacettepe University Faculty of Medicine, Department of Family Medicine; Duygu Ayhan Başer, Assoc. Prof., Study Director — Hacettepe University Faculty of Medicine, Department of Family Medicine; Bahar (Güçiz) Doğan, Prof., Principal Investigator — Hacettepe University Institute of Public Health
Locations (1):
- Hacettepe University Faculty of Medicine, Department of Family Medicine, Family Medicine Training Unit, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No